CLINICAL TRIAL: NCT00360477
Title: Prospective Randomized Trial of Floseal Tubeless Exit vs. Cope Loop Nephrostomy vs. Fascial Stitch Following Percutaneous Nephrolithotripsy
Brief Title: FloSeal Tubeless Exit Versus Cope Loop Nephrostomy Versus Fascial Stitch Following Percutaneous Nephrolithotripsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jaime Landman, Professor and Chairman, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004-3515
Record Dates: First submitted 2006-08-03; First posted 2006-08-04 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Kidney Calculi
Keywords: Kidney stone removal surgery
MeSH Terms: conditions — Kidney Calculi | interventions — FloSeal Matrix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Floseal
  Interventions: Procedure: Floseal
- 2 (Active Comparator): Cope-Loop/Nephrostomy Tube
  Interventions: Procedure: Cope Loop
- 3 (Active Comparator): Fascial Stitch
  Interventions: Procedure: Fascial Stitch

INTERVENTIONS:
Procedure: Floseal — Bioglue that seals the kidney
  Arms: 1
Procedure: Cope Loop — Nephrostomy tube for fluid drainage from the kidney
  Arms: 2
Procedure: Fascial Stitch — Stitch that closes the kidney
  Arms: 3

SUMMARY:
The patient will be asked to participate in a research project designed to determine the best way to prevent bleeding and promote patient comfort after having kidney stones removed. Two standard methods for ending the surgery are being compared to a newer method. In one standard method, the patient will have a tube draining urine from the kidney after the procedure. This tube may also prevent bleeding from the kidney. In another standard method the patient will have a tube left internally that drains urine from the kidney to the bladder and a stitch will be used to close the incision and deeper tissues in the back. In the third potential option, a tube would be left internally to drain urine from the kidney to the patient's bladder and the surgical site would be filled with a clot promoting agent (FloSeal) which is a FDA approved agent specifically formulated to stop bleeding during surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* The patient has kidney stones that require treatment (tx) with percutaneous stone removal
* 18 years of age or over

Exclusion Criteria:

* Patient mentally impaired, have a chronic pain syndrome or disorder, or any condition that might alter the sensation of pain
* Patient taking coumadin
* Pre-existing percutaneous nephrostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-06; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To determine which method of treatment causes the least pain to the patient. | one month

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Louie, MD, Principal Investigator — UC Irvine, Department of Urology
Locations (1):
- University of California, Irvine Medical Center-Department of Urology, Orange, California, United States